CLINICAL TRIAL: NCT05825703
Title: Incidence and Risk Factors of Prolonged Post-Operative Mechanical Ventilation in Pediatric Liver Transplant Recipients: A Retrospective Study
Brief Title: Incidence and Risk Factors of Prolonged Post-Operative Mechanical Ventilation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS/DOA/2022/23757/978
Record Dates: First submitted 2023-04-01; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2022-09

CONDITIONS: Pediatric Liver Transplantation
Keywords: Pediatric Liver Transplantation; Post-operative Mechanical Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PPMV: GROUP OF PATIENT POPULATION WHO HAD PROLONGED POST-OPERATIVE MECHANICAL VENTILATION
- NON PPMV: GROUP OF PATIENT POPULATION WHO DID NOT HAVE PROLONGED POST-OPERATIVE MECHANICAL VENTILATION

SUMMARY:
The primary goal of the study is to identify incidence and risk factors for PPMV in pediatric patients undergoing liver transplantation.

DETAILED DESCRIPTION:
The vast majority of children undergoing orthotopic liver transplantation (OLT) are maintained on mechanical ventilation (MV) in the immediate postoperative period. Reasons for this practice include concerns about graft function, postoperative respiratory depression from opioids, preexisting malnutrition, and organ-recipient size mismatch as well as poor cooperation of young children with postoperative instructions. With current improvements in the perioperative care, there is increasing drive towards early extubation in both adults and children.

Although many children require only a few days of MV following OLT, some require a more prolonged course. In general, prolonged postoperative mechanical ventilation (PPMV) in intensive care unit (ICU) patients is marker of severe adverse events and is associated with higher morbidity and mortality as well as extraordinary resource utilization. Patients requiring PPMV have survived the acute phase of surgery but spend an increased amount of time in the ICU, consume about 50% of all intensive care unit (ICU) resources and are more likely to die. Consequently, investigating the incidence and factors predisposing to PPMV following liver transplant is an important area of research with potential to reduce cost of care and improve long-term outcome of patients.

To our knowledge, factors associated with PPMV following pediatric liver transplantation have not been comprehensively characterized.

ELIGIBILITY:
Inclusion Criteria:

* All Pediatric patients aged <17 years underwent liver transplant between 2010- March 2022 in the institute will be included in the study.

Exclusion Criteria:

* Patients who required mechanical ventilation during the 48 hr preceding surgery.
* Older than 18 yr at the time of transplantation
* Acute liver failure
* Acute on chronic liver failure

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All Pediatric patients aged <17 years underwent liver transplant between 2010- March 2022 in the institute will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-04-30 (Estimated); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with post-operative mechanical ventilation | 24 hours
  To identify risk factors for prolonged post-operative mechanical ventilation (PPMV) in pediatric patients undergoing liver transplantation.

SECONDARY OUTCOMES:
Incidence of PPMV | 24 hours
  To identify risk INCIDENCE for prolonged post-operative mechanical ventilation (PPMV) in pediatric patients undergoing liver transplantation.
total duration of icu stay and length of stay in hospital. | From the day of admission to discharge or death, whichever comes first,upto 12 weeks
  To identify effect of prolonged post-operative mechanical ventilation (PPMV) on total duration of icu stay and length of stay in hospital.
incidence of tracheostomy/re-intubation | 28 days post-op
  To identify incidence of tracheostomy/re-intubation of prolonged post-operative mechanical ventilation (PPMV).
incidence of 28 day mortality | 28 days post-op
  To identify incidence of 28 day mortality prolonged post-operative mechanical ventilation (PPMV) group.

CONTACTS AND LOCATIONS:
Locations (1):
- ILBS, New Delhi, India

IPD SHARING:
Plan to Share IPD: No